CLINICAL TRIAL: NCT02069977
Title: A Multinational, Multicenter, Open-label, Single-arm Study to Evaluate the Efficacy and Safety of Aripiprazole in Asian Pediatric Patients With Autism Spectrum Disorder and Behavior Problems
Brief Title: Study to Evaluate the Efficacy and Safety of Aripiprazole
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yoo-Sook Joung (Other)
Collaborators: Korea Otsuka International Asia Arab (Industry)
Responsible Party: Sponsor-Investigator, Yoo-Sook Joung, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031OTC1301
Record Dates: First submitted 2014-02-13; First posted 2014-02-24 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Autism
Keywords: Autism; Aripiprazole; Abilify
MeSH Terms: conditions — Autistic Disorder | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Experimental): * Dose level: 2, 5, 10, 15 mg/day
  * Starting dose: 2 mg/day
  * Dose increment: The dose should be gradually increased according to the investigator's judgment of subject's response.
  * Target dose: 5-15 mg/day
  * Maximum dose: 15 mg/day
  * Flexibly dosed (2 to 15 mg/day) aripiprazole (oral tablet or solution) is taken once in a day at the same time without regarding to meals
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole
  Other Names: Abilify®

SUMMARY:
* To evaluate the efficacy of flexibly dosed aripiprazole in reducing serious behavioral problems in Asian children and adolescents with a diagnosis of autism spectrum disorder, as measured by change from baseline to endpoint on the irritability subscale of the aberrant behavior checklist (ABC-I).
* To evaluate the long-term safety and tolerability of flexibly dosed aripiprazole in the treatment of serious behavioral problems in Asian children and adolescents with a diagnosis of autism spectrum disorder.

DETAILED DESCRIPTION:
1. Study design

- Multi-national, Multi-center, 52 weeks open label, single arm design

ELIGIBILITY:
Inclusion Criteria:

* 6 to 17 years of age.
* Meeting the diagnostic criteria for autistic disorder specified by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR), with a diagnosis corroborated by the Autism Diagnostic Interview-Revised (ADI-R) diagnostic instrument and demonstrated behaviors such as tantrums, aggression, self-injurious behavior, or a combination of these.
* Clinical Global Impressions (CGI) Severity subscale score ≥ 4 at screening and baseline.
* Aberrant Behavior Checklist (ABC) Irritability subscale score ≥18 at screening and baseline.
* Mental age ≥ 18 months.
* Women of childbearing potential (WOCBP) have to use an adequate method of contraception
* WOCBP must have had a negative serum or urine pregnancy test.
* The patient and/or the designated guardian(s) or caregiver(s) who are able to comprehend and comply with the protocol requirements, in the opinion of the investigator and have consented to participate by signing an informed consent form.

Exclusion Criteria:

* Current diagnosis of bipolar disorder, schizophrenia, major depressive disorder, Rett's disorder, or Fragile-X syndrome.
* History of neuroleptic malignant syndrome.
* Significant risk of committing suicide based on history or routine psychiatric status examination.
* History of seizure in the past 1 year.
* History of severe head trauma or stroke
* History or current evidence of any unstable medical conditions
* Patient considered treatment resistant to neuroleptic medication
* Patient considered treatment resistant to aripiprazole
* Woman who is pregnant or breastfeeding
* ECG: QTc > 475 msec
* Platelets ≤ 75,000/μL
* Hemoglobin ≤ 9 g/dL
* Neutrophils ≤ 1.0x10^3/μL
* Aspartate or alanine transaminase (AST or ALT) > 3xULN
* Serum creatinine ≥ 2 mg/dL
* Patient weighed < 15 kg
* Patient who participated in any other clinical trial within 4 weeks
* Patient determined to require the administration of the prohibited medications during the study period
* Patient with other conditions determined by the investigator to be inappropriate for this clinical study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
irritability subscale of the aberrant behavior checklist | Week 12
  Mean change from baseline to endpoint of Part 1 (week 12)in the caregiver-rated ABC Irritability (ABC-I) subscale score.
  ABC Scale will be completed by subject

SECONDARY OUTCOMES:
Change from baseline in ABC-subscale of lethargy/social withdrawal, stereotypic behavior, hyperactivity, inappropriate speech | Week 1, 2, 4, 8, 12, 24, 36, 52
  ABC Scale will be completed by subject
Change of CGI-S, CGI-I from baseline | Week 1, 2, 4, 8, 12, 24, 36, 52
  CGI-S, CGI-I scale will be evaluated by investigator
Change of Behavioral problems from baseline | Week 12, 52
  Behavioral problems scale: Child Yale-Brown Obsessive-Compulsive Scale (CY-BOCS)
Change of Adaptive Skills from baseline | week 12, 52
  Adaptive Skills Scale: Vineland Adaptive Behavior Scale (VABS)
Change of Parental stress from baseline | Weekk 12, 52
  Parental stress scale: Parenting Stress Index (PSI)

OTHER OUTCOMES:
Adverse events (AEs) | Week 1, 2, 4, 8, 12, 24, 36, 52
  Safety will be evaluated based on below inormaiton.
  * Laboratory test results (routine lab. and serum prolactin)
  * Vital signs (blood pressure, pulse, body temperature)
  * ECG
  * Weight gain
  * Extrapyramidal side effects (EPSEs) assessed by Simpson-Angus Rating Scale (SAS), Barnes Akathisia Rating Scale (BARS), and Abnormal Involuntary Movement Scale (AIMS)

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-Sook Joung, MD. PhD., Principal Investigator — Sumsung Medical Center
Locations (6):
- Philippines (2):
  - Medical City, Pasig
  - Philippine Children's Medical Center, Quezon City
- South Korea (3):
  - Inje University Ilsan Paik Hospital, Ilsan, Gyeonggi-do
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Siriraj Hospital Mahidol University, Bangkok, Thailand

REFERENCES:
- [Derived] Kim BU, Kim HW, Park EJ, Kim JH, Boon-Yasidhi V, Tarugsa J, Reyes A, Manalo SG, Joung YS. Long-Term Improvement and Safety of Aripiprazole for Irritability and Adaptive Function in Asian Children and Adolescents with Autistic Disorder: A 52-Week, Multinational, Multicenter, Open-Label Study. J Child Adolesc Psychopharmacol. 2022 Sep;32(7):390-399. doi: 10.1089/cap.2022.0004. PMID 36112116